CLINICAL TRIAL: NCT04643600
Title: The Effect of Orally Administered L- Arginine on Quadriceps Strenght in Healthy Smokers
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Goranka Radmilović (Other)
Responsible Party: Sponsor-Investigator, Goranka Radmilović, physiatrist, principal investigator, Daruvarske Toplice
Organization: Daruvarske Toplice (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: 2156-61-07-20-170
Record Dates: First submitted 2020-11-19; First posted 2020-11-25 (Actual); Last update posted 2021-08-23 (Actual); Status verified 2021-08

CONDITIONS: Spirometry; Qadriceps Muscle
Keywords: COPD; L-arginine; locomotor parameters; smokers; quadriceps muscle
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Arginine

STUDY DESIGN:
Intervention Model Description: The research will be organized as a cross-sectional study that will include patients, smokers and non-smokers, who are undergoing medical rehabilitation or medically programmed vacation in the Special Hospital for Medical Rehabilitation Daruvarske toplice
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Smokers (Active Comparator): The strength test of the the quadriceps muscle, will be measured in all patients on the Biodex isokinetic device. Quadriceps strength testing will be performed on 2 occasions. On one occasion without medication, except those that the patient may take permanently, and on the other 90 minutes after the patient takes 1 tbl of L - Arginine 500 mg on mouth to an empty stomach ,in order to monitor the possible increase in quadriceps strength. All patients who are smokers will have recorded : the age of onset of smoking, the year of smoking experience and the average number of cigarettes smoked per day. All patients will complete the CAT, IPAQ and DASS-21 questionnaire.
  Interventions: Drug: L-Arginine, 500 Mg Oral Capsule
- Non - smokers (Active Comparator): All patients will be maesured: body weight, height, BMI (body mass index), waist circumference, pulse (cp), saturation (SpO2), blood pressure, respiratory index and thoracic spine mobility index measured. All patients will do a 6-minute walk test and test on a bicycle erogometer. The strength test of the the quadriceps muscle, will be measured in all patients on the Biodex isokinetic device. Quadriceps strength testing will be performed on 2 occasions. On one occasion without medication, except those that the patient may take permanently, and on the other 90 minutes after the patient takes 1 tbl of L - Arginine 500 mg on mouth to an empty stomach ,in order to monitor the possible increase in quadriceps strength. All patients will complete the CAT, IPAQ and DASS-21 questionnaire.
  Interventions: Drug: L-Arginine, 500 Mg Oral Capsule

INTERVENTIONS:
Drug: L-Arginine, 500 Mg Oral Capsule — The strength test of the the quadriceps muscle, will be measured in all patients on the Biodex isokinetic device. Quadriceps strength testing will be performed on 2 occasions. On one occasion without medication, except those that the patient may take permanently, and on the other 90 minutes after the patient takes 1 tbl of L - Arginine 500 mg on mouth to an empty stomach ,in order to monitor the possible increase in quadriceps strength.

SUMMARY:
The study will investigate changes in certain locomotor parameters as early predictors of disease in smokers who are prone to develop chronic obstructive pulmonary disease (COPD).

DETAILED DESCRIPTION:
The research will include about 150 respondents aged 40-65, smokers and non-smokers, and will be conducted at the Special Hospital for Medical Rehabilitation 'Daruvarske toplice'. All patients will make spirometry and the Tiffeneau-Pinelli index (ratio of forced expiratory volume in 1 second - FEV1 and forced vital capacity FVC).

All patients will be maesured: body weight, height, BMI (body mass index), waist circumference, pulse (cp), saturation (SpO2), blood pressure, respiratory index and thoracic spine mobility index measured. The thickness of the skin fold will be measured on the abdomen with a caliper and on the measuring device for the analysis of body mass composition - Gaia, the percentage of muscle and fat tissue will be determined for each patient, as well as the analysis of body mass composition. All patients will do a 6-minute walk test and the patient's cardiorespiratory and muscular ability will be tested on a bicycle erogometer, the values of maximal oxygen uptake (VO2 max) and pulse (cp) will be recorded and the patient's fitness status determined. Each patient will estimate dyspnea intensity from 1 -10 before and after a 6-minute walk test and before and after a bicycle ergometer according to the Borg's dyspnea scale. The strength test of the the quadriceps muscle, will be measured in all patients on the Biodex isokinetic device. Quadriceps strength testing will be performed on 2 occasions. On one occasion without medication, except those that the patient may take permanently, and on the other 90 minutes after the patient takes 1 tbl of L - Arginine 500 mg on mouth to an empty stomach ,in order to monitor the possible increase in quadriceps strength. All patients who are smokers will have recorded : the age of onset of smoking, the year of smoking experience and the average number of cigarettes smoked per day. All patients will complete the CAT, IPAQ and DASS-21 questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* aged 40-65
* smokers and non-smokers, All patients will make spirometry and the Tiffeneau-Pinelli index (ratio of forced expiratory volume in 1 second - FEV1 and forced vital capacity FVC)> 75% of the predictive value will be taken as an inclusion criteria.

Exclusion Criteria:

* FEV1 / FVC <75%,
* inflammatory rheumatic diseases,
* malignancies,
* acute and severe heart or lung disease,
* unregulated hypertension,
* patients who have undergone major surgery in the past year,
* patients with implanted hip, knee or ankle prosthesis, will be excluded from the study.

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 163 (Estimated)
Dates: Start 2019-03-01 (Actual); Primary Completion 2022-02-15 (Estimated); Study Completion 2022-02-17 (Estimated)

PRIMARY OUTCOMES:
Quadriceps strenght | 1 day between two tests, 90min after taking L- Arginine a 500mg
  Quadriceps strength testing will be performed on 2 occasions. On one occasion without medication, except those that the patient may take permanently, and on the other 90 minutes after the patient takes 1 tbl of L - Arginine 500 mg on mouth to an empty stomach ,in order to monitor the possible change in quadriceps strength.

CONTACTS AND LOCATIONS:
Locations (1):
- Daruvarske Toplice, Daruvar, Bjelovar-Bilogora County, Croatia

IPD SHARING:
Plan to Share IPD: No